CLINICAL TRIAL: NCT00984789
Title: Transdermal Contraception Patch: EU Cycle Control Study Versus EVRA
Brief Title: Birth Control Patch Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13082; 2008-007308-27 (EudraCT Number)
Record Dates: First submitted 2009-09-04; First posted 2009-09-25 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Contraception
Keywords: Transdermal Patch; Bleeding; Pregnancy
MeSH Terms: conditions — Hemorrhage | interventions — Ethinyl Estradiol; Gestodene; norelgestromin; Ortho Evra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Ethinylestradiol/Gestodene (FC Patch Low BAY86-5016)
- Arm 2 (Active Comparator)
  Interventions: Drug: Norelgestromin/Ethinylestradiol (EVRA)

INTERVENTIONS:
Drug: Ethinylestradiol/Gestodene (FC Patch Low BAY86-5016) — 0.55mg ethinylestradiol and 2.1mg gestodene
  Arms: Arm 1
Drug: Norelgestromin/Ethinylestradiol (EVRA) — 0.6mg ethinylestradiol and 6mg norelgestromin
  Arms: Arm 2

SUMMARY:
400 healthy women needed contraception will be asked to participate in this study. Half will be given EVRA, half will be given FC Patch low. They will be expected to apply the patches for 21 days of their cycle, for 7 cycles in total. The study will compare the patterns of menstrual bleeding on these two treatments, plus how effective they are at preventing pregnancy, general safety, and their acceptability to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women requesting contraception aged 18-35 years old
* Smokers must not be older than 30 at time of informed consent
* History of regular cyclic menstrual periods, normal cervical smear

Exclusion Criteria:

* Pregnancy or lactation
* Obesity (BMI>30), hypersensitivity to any ingredients of the study drug, significant skin reaction to transdermal preparations, any diseases/conditions that can compromise the functions of the body system (resulting in altered absorption/accumulation/ metabolism/excretion of the study drug), any diseases / conditions that may worsen under hormonal treatment

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 393 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Bleeding Patterns and cycle control | 7 cycles (each consisting of 28 days)

SECONDARY OUTCOMES:
Contraceptive efficacy | 7 cycles (each consisting of 28 days) + follow up period of 14 days
Adverse Event Collection | 7 cycles (each consisting of 28 days)
Population pharmacokinetics | 7 cycles (each consisting of 28 days)
Compliance to treatment | 7 cycles (each consisting of 28 days)
Subjective assessment of treatment | 7 cycles (each consisting of 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- Austria (9):
  - Mödling, Lower Austria
  - Wiener Neustadt, Lower Austria
  - Graz, Styria
  - Wörgl, Tyrol
  - Bregenz, Vorarlberg
  - Graz
  - Innsbruck
  - Vienna
  - Zeltweg
- Czechia (6):
  - Brno
  - České Budějovice
  - Hradec Králové
  - Olomouc
  - Písek
  - Prague
- Netherlands (4):
  - De Bilt
  - Den Helder
  - Heerlen
  - Nijmegen

REFERENCES:
- [Derived] Gruber D, Skrivanek A, Serrani M, Lanius V, Merz M. A comparison of bleeding patterns and cycle control using two transdermal contraceptive systems: a multicenter, open-label, randomized study. Contraception. 2015 Feb;91(2):105-12. doi: 10.1016/j.contraception.2014.10.003. Epub 2014 Oct 13. PMID 25453582